CLINICAL TRIAL: NCT05649956
Title: A Randomized Phase II Study of Letrozole Versus Observation in Patients with Newly Diagnosed Uterine Leiomyosarcoma
Brief Title: Letrozole in Uterine Leiomyosarcoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: GOG Foundation (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GOG-3088
Record Dates: First submitted 2022-12-06; First posted 2022-12-14 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Uterine Leiomyosarcoma
MeSH Terms: interventions — Letrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Letrozole (Experimental): Letrozole 2.5 mg orally
  Interventions: Drug: Letrozole
- Observation (No Intervention): Observation

INTERVENTIONS:
Drug: Letrozole — Letrozole 2.5 mg PO daily
  Arms: Letrozole

SUMMARY:
This is a clinical trial to test letrozole in patients with uterine leiomyosarcoma. The main question is will treatment with letrozole extend progression-free survival in patients. Patients will receive 2/5 mg of letrozole daily.

DETAILED DESCRIPTION:
This is a randomized phase II study of letrozole (Femara) administered 2.5 mg orally daily to patients with newly diagnosed clinical stage I and II LMS. Using an adaptive randomization, patients will be assigned to either the treatment arm (letrozole group) or observation. The primary outcome for this trial is the time to progression.

ELIGIBILITY:
Inclusion Criteria:

1. Patient or a legally authorized representative must have signed an approved informed consent and authorization permitting the release of personal health information.
2. Patient must have histologically confirmed newly diagnosed uterine leiomyosarcoma with disease limited to the uterus (FIGO 2009 Stage I). Submission of pathology report documenting uterine leiomyosarcoma histology is required in the IRT Source Document Portal following randomization.
3. Patient tumors must express ER positivity by immunohistochemistry (ER expression greater than 10% by immunohistochemistry). ER status test results must be provided at enrollment. Sites are required to report results of ER status testing in the IRT Source Document Portal.
4. Patient must have completed hysterectomy and bilateral salpingo-oopherectomy no more than 12 weeks from enrollment.
5. All patients must have NO measurable disease as defined by RECIST 1.1 within 6 weeks of enrollment. Measurable disease is defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded). Each lesion must be greater than or equal to 10 mm when measured by CT, MRI or caliper measurement by clinical exam; or greater than or equal to 20 mm when measured by chest x-ray. Lymph nodes must be greater than or equal to 15 mm in short axis when measured by CT or MRI.
6. Patients must have an ECOG performance status of 0, 1, or 2.
7. Patients must have adequate organ and marrow function as defined below:

   NOTE: Institutional/laboratory upper limit of normal = ULN Institutional/laboratory lower limit of normal = LLN

   Bone marrow function:
   * Absolute neutrophil count (ANC) greater than or equal to 1500 cells/mcl
   * Platelet count greater than or equal to 100,000 cells/mcl
   * Hemoglobin greater than or equal to 9.0 g/dL (Patients may receive erythrocyte transfusions to achieve this hemoglobin level at the discretion of the Investigator. Initial treatment must not begin earlier than the day after erythrocyte transfusion).

   Renal function:

   • Serum creatinine less than or equal to 1.5 x ULN

   Hepatic function:
   * AST (aspartate aminotransferase) and ALT (alanine aminotransferase) less than or equal to 3.0 x ULN
   * Serum albumin greater than or equal to 2.5 g/dL
8. Patient must be at least 18 years of age.
9. Patient must be able to swallow oral medication.

Exclusion Criteria:

Exclusion Criteria 1. Patients who do not have pure uterine sarcomas (i.e., no mixed malignant mullerian tumors are permitted).

2. Patients with any other severe concurrent disease, which would make the patient inappropriate for entry into this study, including significant hepatic, renal, or gastrointestinal diseases.

3. Patients with concomitant invasive malignancy or a history of prior malignancy except non-melanoma skin cancer, in situ cervical cancer, or other cancer for which the patient has been disease-free for at least three years. Patients are also excluded if their previous cancer treatment contraindicates this protocol.

4. Patients who have a history of taking any aromatase inhibitor within the past 5 years.

5. Patients with active or uncontrolled systemic infection. 6. Patients with history of uncontrolled cardiac disease, i.e., uncontrolled hypertension (defined as systolic greater than 150 mm Hg or diastolic greater than 90 mm HR despite antihypertensive medications), unstable angina, recent myocardial infarction (within prior 6 months), uncontrolled congestive heart failure (NYHA Class II or greater), clinically significant cardiac arrhythmias, and cardiomyopathy with an ejection fraction under 40%.

7. Patients currently receiving chemotherapy or radiation therapy. 8. Patients with severe hepatic impairment and/or cirrhosis. 9. Patients with duodenal stent or other GI disorder/defect that would interfere with absorption of oral medication.

10. Patients deemed otherwise clinically unfit for clinical trial per investigators discretion.

11. Patients with known hypersensitivity to any of the excipients of letrozole. 12. Patients who are pregnant or breast-feeding. 13. Patients who are currently part of or have participated in any clinical investigation with an investigational drug within 30 days of prior to enrollment.

14. Patients currently using systemic estrogens, including herbals and supplements with estrogenic properties. The use of vaginal estrogen is permitted if symptoms are refractory to moisturizers and lubricants.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 40 (Estimated)
Dates: Start 2024-07-17 (Actual); Primary Completion 2028-07-30 (Estimated); Study Completion 2029-07-30 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | Measured from time of enrollment until date of progression or death up 3 years from randomization

CONTACTS AND LOCATIONS:
Overall Officials: Bradley Corr, MD, Study Chair — University of Colorado, Denver
Locations (12):
- United States (12):
  - University of Colorado Cancer Center - Anschutz Cancer Pavilion, Aurora, Colorado
  - Highlands Ranch Hospital, Highlands Ranch, Colorado
  - Mount Sinai Comprehensive Cancer Center, Miami Beach, Florida
  - Endeavor Health - Kellogg Cancer Center, Evanston, Illinois
  - WK Physician Network-Gynecologic Oncology Associates, Shreveport, Louisiana
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - Women's Cancer Center of Nevada, Las Vegas, Nevada
  - University of New Mexico Comprehensive Cancer Center, Albuquerque, New Mexico
  - East Carolina University Health Medical Center, Greenville, North Carolina
  - University of Oklahoma Health Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Asplundh Cancer Pavilion, Willow Grove, Pennsylvania
  - Woman and Infants Hospital of Rhode Island, Providence, Rhode Island

IPD SHARING:
Plan to Share IPD: No